CLINICAL TRIAL: NCT03522961
Title: Cranberry Tablets Versus Nitrofurantoin Prophylaxis for Urinary Tract Infection Prevention After Urogynecologic Surgery: a Double-blinded Randomized Clinical Trial
Brief Title: Cranberry Tablets Versus Nitrofurantoin Prophylaxis for Urinary Tract Infection Prevention After Urogynecologic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Theralogix LLC (Unknown)
Responsible Party: Principal Investigator, Jeannine Marie Miranne, Urogynecologist; Assistant Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017P002904; 016086 (Other Grant/Funding Number: Brigham and Women's Hospital OB/GYN Department)
Record Dates: First submitted 2018-04-17; First posted 2018-05-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Urinary Tract Infections; Pelvic Organ Prolapse; Urinary Incontinence
MeSH Terms: conditions — Urinary Tract Infections; Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrofurantoin prophylaxis/Placebo (Active Comparator): Subjects will receive Nitrofurantoin 100mg capsules (Bottle A) once a day until they pass their voiding trial and no longer require transurethral catheterization. Subjects will be switched to Placebo capsules (Bottle B) once a day, starting the day after they pass their voiding trial until the end of the 28 day study period.
  Interventions: Drug: Nitrofurantoin Prophylaxis/Placebo
- Cranberry capsules (Active Comparator): Subjects will receive TheraCran® One Cranberry 36mg capsules (Bottle A) once a day until they pass their voiding trial and no longer require transurethral catheterization. Subjects will be switched to another bottle of TheraCran® One Cranberry 36mg capsules (Bottle B) once a day, starting the day after they pass their voiding trial until the end of the 28 day study period.
  Interventions: Drug: Cranberry capsules

INTERVENTIONS:
Drug: Nitrofurantoin Prophylaxis/Placebo — Drug: Nitrofurantoin Drug: Placebo
  Arms: Nitrofurantoin prophylaxis/Placebo
Drug: Cranberry capsules — Drug: TheraCran® One Cranberry capsules
  Arms: Cranberry capsules

SUMMARY:
We aim to compare the effectiveness of cranberry capsules versus nitrofurantoin prophylaxis in preventing urinary tract infections (UTIs) after urogynecologic surgery by conducting a double-blinded randomized clinical trial involving women with pelvic organ prolapse and/or urinary incontinence scheduled to have surgery with the Urogynecologists who comprise the Brigham and Women's Urogynecology Group.

DETAILED DESCRIPTION:
We plan to conduct a double-blinded randomized clinical trial involving women who undergo surgery for pelvic organ prolapse and/or urinary incontinence.

Participants who need transurethral catheterization postoperatively will be randomized to cranberry capsules or nitrofurantoin prophylaxis. Randomization will be performed the day of discharge. Both participants and surgeons will be blinded to treatment allocation. All participants will receive routine perioperative intravenous antibiotic prophylaxis.

Participants who fail their voiding trial after surgery and require transurethral catheterization upon discharge from the hospital will be randomized to either one cranberry capsule (TheraCran one®, Theralogix, LLC, Rockville, Maryland) or one 100 mg capsule of nitrofurantoin by mouth daily beginning postoperative day #1. Participants randomized to the cranberry capsule group will continue to take one cranberry capsule daily for 28 days. Participants randomized to the nitrofurantoin group will continue to take 100 mg of nitrofurantoin each day transurethral catheterization is needed for up to 28 days. All participants will be scheduled for a repeat voiding trial within 48 hours to 1 week after discharge.

All participants will complete a daily catheterization and medication diary to record the type of catheterization used (indwelling or intermittent) and to confirm they are taking the study medication for the duration of the study period. They will also be asked to record any urinary symptoms they experience and will be encouraged to contact the office immediately if they experience urinary symptoms consistent with a UTI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* English-speaking
* Plan for pelvic organ prolapse (POP) or urinary incontinence (UI) surgery

Exclusion Criteria:

* Pregnancy
* Urethral diverticulectomy
* Urogenital fistula repair
* Sacral neuromodulation
* Congenital urogenital anomaly
* Allergy to cranberry products
* Allergy to nitrofurantoin
* Dependent on catheterization preoperatively
* Recurrent UTI's (3 or more culture proven UTI's over the past consecutive 12 months)
* Known creatinine clearance <60 mL/min
* Non-English, Non-Spanish speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be treatment for clinically suspected or culture-proven UTI in the cranberry capsule group versus the nitrofurantoin group within 4 weeks (28 days) after surgery. | 28 days
  Clinically suspected treatment will include both empiric treatment based on the development of urinary symptoms alone (dysuria, urinary urgency, and/or urinary frequency) or prescribed based on symptoms suggestive of a UTI and the presence of nitrites and/or leukocyte esterase on urine dipstick analysis. Participants will fill out a daily catheterization and medication diary which asks about the presence or absence of UTI symptoms. They will be encouraged to call the office and/or come in for evaluation if they experience these symptoms. These participants may be treated based on their symptoms alone or based on their symptoms and the presence of nitrites and/or leukocyte esterase on urine dipstick analysis. A culture-proven UTI will be defined as a urine culture result with >100,000 colony-forming units of a single organism.

SECONDARY OUTCOMES:
Prevalence of bacterial resistance to nitrofurantoin on postoperative urine cultures for those participants who have culture-proven UTIs | 28 days
Adherence to assigned treatment:cranberry capsule vs. nitrofurantoin | 28 days
  A daily catheterization and medication diary will be used to track whether or not participants took their study medication every day for 28 days. Participants will bring their study medication bottle to every study visit and the medication will be counted by study staff to ensure adherence to assigned treatment.
Reasons for non-adherence to assigned treatment | 28 days
  At office visits throughout the study period, after the participants' study medication is counted and non-adherence to assigned treatment is found, study physicians will ask participants for their reasons for non-adherence.
Risk factors for postoperative UTI | 28 days
  Risk factors for postoperative UTI will be assessed based on the participants' individual medical history and physical exam. Risk factors will be assessed by study physicians at office visits throughout the study period.
Time to first postoperative UTI | 28 days
Number of postoperative UTIs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeannine M Miranne, MD, MS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No